CLINICAL TRIAL: NCT06883747
Title: A Phase 0/1 Study of BMS-986504, a MTA Cooperative PRMT5 Inhibitor in Recurrent Glioblastoma Participants With MTAP Deleted Tumors Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration With PK-Triggered Expansion Cohort
Brief Title: Clinical Trial of BMS-986504 in Recurrent GBM Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Responsible Party: Sponsor-Investigator, Nader Sanai, Director, Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-21
Record Dates: First submitted 2025-02-25; First posted 2025-03-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma WHO Grade IV
Keywords: MTAP loss; MTAP deletion; MTAP del

STUDY DESIGN:
Intervention Model Description: Single dose escalation arm with 3 dose cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recurrent WHO Grade 4 Glioblastoma MTAP loss/deletion (Experimental)
  Interventions: Drug: BMS-986504

INTERVENTIONS:
Drug: BMS-986504 — MTA cooperative PRMT5 inhibitor
  Other Names: MRTX1719

SUMMARY:
This is an open-label, multi-center, Phase 0/1 dose-escalation trial designed to enroll up to 9 total recurrent glioblastoma (rGBM) participants with confirmed MTAP loss/deletion in their archival or pretreatment biopsy tissue, who are scheduled for surgical resection. MTAP loss/deletion will be determined by next-generation sequencing (NGS). The trial will include a dose escalation design to evaluate the pharmacokinetics (PK) and safety and tolerability of BMS-986504 (MRTX1719). The trial will be composed of a Phase 0 component and an Expansion Phase 1 component. Participants with tumors demonstrating a positive PK response in the Phase 0 component of the study will be eligible to enroll into the the Phase 1 component that will include 21-day cycles of therapeutic dosing of BMS-986504.

DETAILED DESCRIPTION:
PHASE 0

Eligible participants will enroll in the Phase 0 study and receive BMS-986504 in three dose escalation cohorts over 6 days prior to surgical resection. The final dose will be administered 3-5 hours before tumor resection on Day 6. Participants without histologically confirmed diagnosis of recurrent GBM after the craniotomy will be replaced.

Phase 0 Dose Escalation

An initial cohort of three participants will be enrolled at the starting dose level. If ≤1 of the participants experiences a dose-limiting toxicity (DLT) through the end of the Phase 0, the dose is escalated to the next level. Dose escalation continues to the next level if no more than one out of three participants experience a DLT. However, if two or more participants experience DLTs at any dose level, dose escalation stops.

A written report will be submitted to the DSMB Chair (or qualified alternate) describing the time intervals, dose levels, adverse events, safety reports and any DLTs observed after enrollment into each cohort is complete. The DSMB Chair will review the report and provide a written authorization to proceed or will request more information within approximately 2 business days. Approval for the initiation of enrollment must be obtained prior to implementation.

Phase 0 Dose Limiting Toxicity (DLT)

DLTs will be defined as any adverse event that is not clearly due to the underlying disease or extraneous causes, t and unrelated to disease, disease progression, intercurrent illness or concomitant medications from Phase 0 Day 1 through termination from the study or study completion. DLTs will include:

* ≥ Grade 3 thrombocytopenia with clinically significant bleeding
* > Grade 4 neutropenia for more than 7 days
* Neutropenic fever
* As determined by the investigator, any unacceptable toxicity which may include treatment-related death or grade 4 toxicity
* Any non-hematologic toxicity:

  * Grade ≥ 3 regardless of relatedness to study treatment, duration, or baseline grade;
  * Events that meet Hy's law criteria;
  * Excluding the following:

    * Grade 3 nausea/vomiting or diarrhea for less than 72 hours with adequate antiemetic and other supportive care
    * Grade 3 fatigue for greater than 1 week
    * Grade 3 or higher electrolyte abnormality that lasts up to 72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional medical interventions
* Any death not clearly due to the underlying disease or extraneous causes

Phase 0 PK/PD Assessments Tumor PK and PD analyses will be performed at IVY. To assess the PK and PD endpoints listed, blood, CSF and brain tumor tissue (Gd-enhancing and Gd-non-enhancing tumor tissue will be collected and analyzed separately) will be collected intraoperatively.

Retrospective genomic analysis of tissue from Phase 0 and subsequent resections at recurrence will be performed if positive PK/PD responses are observed.

Participants with tumors demonstrating negative PK will not proceed to the Expansion Phase 1 component but will receive standard of care. Participants will complete the end-of-treatment visit, safety follow-up, and survival monitoring as outlined in the "All Participants" section.

PHASE 1

Participants with tumors demonstrating PK response will continue treatment with the same dose that was received in Phase 0 once daily (QD) in a continuous regimen expressed in 3-week (21-day) cycles. Treatment will begin once the participant has recovered from surgery. Participants will receive BMS-986504 until the progression of disease, unacceptable toxicity or death, withdrawal of consent, loss to follow-up, or study termination by sponsor. Participants will complete the end-of-treatment visit, safety follow-up, and survival monitoring as outlined in the "All Participants" section.

Phase 1 Dose Modifications

Participants who experience a clinically significant Grade 2 toxicity considered related to study treatment, or a Grade 3 or 4 toxicity considered related to study treatment may temporarily suspend study treatment. Depending on the toxicity, study treatment may resume within 28 days after discussion with the Safety Officer.

Dosing of BMS-986504 during Phase 1 can be interrupted for approximately 28 days for medical events that are not associated with toxicity related to study treatment or disease progression.

Criteria for treatment modifications and suggested guidelines for the management of toxicities related to BMS-986504 are summarized in the protocol. These general guidelines may be modified at the discretion of the Investigator based on the best clinical judgement at that time. Any toxicities related to BMS-986504 should be managed according to standard medical practice.

A participant must discontinue study treatment, if, after treatment is resumed at a lower dose, the toxicity recurs with the same or worse severity.

ALL PARTICIPANTS

All participants will return to the clinic for safety monitoring per the schedule of activities following treatment discontinuation and will be contacted approximately every 3 months for up to 12 months for survival data collection. MRI scans and review to monitor progression in guidance with RANO criteria will occur approximately 2-3 month, per standard of care. The start of follow-up for long-term survival begins following completion of the Day 30 safety follow up call.

At treating physician's discretion, longitudinal biomarker analysis through liquid biopsy will be conducted to characterize genomic and/or transcriptomic changes from tumor cells or cell-free DNA collected from CSF at Phase 0, at Expansion Phase, or recurrent craniotomy.

Additional biomarker analysis may be conducted using surgical tissue. If the participant undergoes repeat craniotomy for recurrence or progression of his/her brain tumor, IVY will request samples from the resected tumor, CSF or blood to enable longitudinal sample collection and analysis that will help identify possible resistance mechanisms.

STUDY STOPPING CRITERIA

Study stopping rules are:

* If < 1 of 3 participant shows positive PK at the highest dose level.
* If ≥ 2 participants have a ≥ 4-week delay to surgery due to BMS-986504 related toxicity at any dose level.
* Any unacceptable toxicity such as Grade 4 toxicity or death not clearly related to underlying disease or extraneous cause

The following options may occur as a result of any of the above:

* Halt participant dosing or study enrollment until the toxicity data can be further studied by the DSMB.
* Amend the protocol to address any of the below:

  * Evaluate additional subjects in a particular dose cohort or in each dose cohort to make the study more sensitive to characterizing adverse events;
  * Implementation of smaller dose increases between dose cohorts;
  * Exclusion of certain participants thought to be more at-risk for a particular adverse event.
* Stop the study.

STUDY OBJECTIVES The Phase 0 Primary Objective is to evaluate concentration of BMS-986504 in Gd-non-enhancing tumor tissue, and the Expansion Phase Primary Objective is to assess safety and tolerability of BMS-986504 in participants who receive at least one dose.

The Phase 0 Secondary Objective is to evaluate concentration of BMS-986504 in CSF collected during Phase 0 surgery, and the Expansion Phase Secondary Objectives are to measure the rate of 6-month progression free survival (PFS6) and examine overall survival (OS) in participants.

STUDY DURATION The estimated total study length of around 15 months includes study initiation and accrual of 9 participants in 9 months, and follow-up for the participants for an additional 6 months to conclude the study.

The final trial report will be summarized and submitted for peer-review journals for publication

Phase 0 Participants: Up to approximately 2 months (screening window of 28 days through Day 30 phone call follow-up).

Phase 1 Participants: BMS-98604 will be taken by the participant as long as the drug is tolerated, and the investigator believes the participant may be obtaining benefit. Treatment will be taken by the participant until confirmed progression, unacceptable toxicity, death, withdrawal of consent, lost to follow-up, or end of treatment.

All Participants: Participants will be followed for survival for up to 12 months following end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the diagnosis of glioblastoma by the 2021 WHO criteria, who have progressed on or following previous tumor-directed therapy, which must have included a maximal safe resection (biopsy allowed if it was deemed unsafe to resect) and fractionated radiotherapy (RT).
* Patients with archival tissue demonstrating MTAP loss/deletion confirmed through NGS will be qualified for Phase 0 portion of the study.
* Participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm.
* Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤ 1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Day 1. A washout period of at least 21 days is required between the last chemotherapy dose and Day 1 (provided the participant did not receive RT).
* Age ≥ 18 at time of consent
* Have a performance status (PS) of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

  * Adequate Bone Marrow Function: Absolute neutrophil count ≥ 1,500/mcL; Platelets (at time of surgery) ≥ 100,000/mcL; Hemoglobin ≥ 9.0 g/dL (participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)
  * Adequate Hepatic Function: Total Bilirubin ≤ 1.5 X ULN; Participants with Gilbert's syndrome with a total bilirubin ≤ 2.0 times ULN and direct bilirubin within normal limits are permitted; AST (SGOT) ≤ 3 X institutional ULN; ALT (SGPT) ≤ 3 X institutional ULN
  * Adequate Renal Function: Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2 by Chronic Disease Epidemiology Collaboration (CKD-EPI) equation; Serum creatinine ≤ 1.5 X ULN or estimated creatinine clearance >/= 60 mL/min (calculated using Institutional standard method)
  * Coagulation Function: INR ≤ 1.5 X ULN
* Ability to swallow oral medications without crushing or chewing.
* Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
* For females of reproductive potential: use of highly effective contraception for at least 28 days prior to treatment and agreement to use such a method during study participation and for an additional 7 months after the end of treatment administration.
* Females of child-bearing potential must agree not to breastfeed starting at screening, throughout the study period and for 7 months after final study drug administration.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and avoid sperm donation for the duration of the study and for an additional 4 months after the end of treatment administration.
* Agreement to adhere to Lifestyle Considerations throughout study duration.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
* Participant understands the informed consent document and has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative(s), and assent if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.

Exclusion Criteria:

* Inability to undergo MRI brain with intravenous (IV) contrast
* Known active systemic bacterial infection (IV antibiotics or fever > 38.5°C at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening of viral infection is not required for enrollment.
* Cardiovascular abnormalities including:

  * LVEF < 50%
  * History of prolonged QTc, or QT interval corrected for heart rate using Fridericia's formula (QTcF) prolongation > 480 msec, except for right bundle branch block.
  * Uncontrolled/symptomatic or significant cardiovascular conditions within 6 months prior to enrollment, including but not limited to any of the following: Cardiac angioplasty or stenting, unstable angina pectoris, myocardial infarction, stroke/transient ischemic attack, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, New York Heart Association (NYHA) class III-IV congestive heart failure, pericarditis, atrial fibrillation or other arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes).
* Symptomatic or radiographic leptomeningeal disease.
* Known other concurrent severe and/or uncontrolled medical condition that, in the investigator's judgment, would cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g., Celiac disease, Crohn's disease, gastric bypass, malabsorption, chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) Grade 1 at the time of starting study treatment and patients with chronic Grade 2 unresolved toxicities may be eligible following discussion with the Principal Investigator.
* Treatment with another investigational drug or other intervention within 5 half-lives of the investigational product whichever is longer.
* Prior treatment with another PRMT5 inhibitor.
* Known allergic reactions to components of BMS-986504: microcrystalline cellulose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol/macrogol, and talc.
* Use of strong inhibitors and strong inducers of CYP3A4/P-gp. Consider using alternative medications, per Investigator judgment.
* Concurrent use of medications known to prolong the QT interval (e.g., certain antiarrhythmics, antibiotics, antipsychotics, and antidepressants) unless discontinued for an appropriate washout period as determined by the investigator.
* Participants who have received live/attenuated vaccine within 30 days of anticipated first treatment. The use of inactivated seasonal influenza vaccines (e.g., Fluzone®) will be permitted on study without restriction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
BMS-986504 Concentration in Tumor Tissue | intraoperative
  Total and unbound BMS-986504 concentration will be quantified in Gd-enhancing and Gd-non-enhancing tumor tissue collected during Phase 0 surgery.
Number of Treatment-Emergent Adverse Events | From date of enrollment until 30 days after last dose, assessed over 15 months
  Safety and tolerability of BMS-986504 will be assessed by tabulating (Number and Percent) Treatment-Emergent Adverse Events (TEAEs) according to the highest grade observed per participant for each event or category (per CTCAE v5.0). The analysis population includes participants who took at least one dose of the study drug.
Number of Treatment-Related Adverse Events | From date of first dose of study drug until 30 days after last dose, assessed over 15 months
  Safety and tolerability of BMS-986504 will be assessed by tabulating (Number and Percent) Treatment-Related Adverse Events (TEAEs) according to the highest grade observed per participant for each event or category (per CTCAE v5.0). The analysis population includes participants who took at least one dose of the study drug.
Number of Serious Adverse Events | From date of enrollment until 30 days after last dose, assessed over 15 months
  Safety and tolerability of BMS-986504 will be assessed by tabulating (Number and Percent) Serious Adverse Events (SAEs) according to the highest grade observed per participant for each event or category (per CTCAE v5.0). The analysis population includes participants who took at least one dose of the study drug.
Number of Clinical Laboratory Abnormalities | From date of enrollment until 30 days after last dose, assessed over 15 months
  Safety and tolerability of BMS-986504 will be assessed by tabulating (Number and Percent) Clinical Laboratory Abnormalities according to the highest grade observed per participant for each event or category (per CTCAE v5.0). The analysis population includes participants who took at least one dose of the study drug.
Number of Drug-Related Toxicities | From date of first dose of study drug until 30 days after last dose, assessed over 15 months
  Safety and tolerability of BMS-986504 will be assessed by tabulating (Number and Percent) Drug-Related Toxicities (defined by Dose Limiting Toxicities) according to the highest grade observed per participant for each event or category (per CTCAE v5.0). The analysis population includes participants who took at least one dose of the study drug.

SECONDARY OUTCOMES:
BMS-986504 Concentration in Cerebrospinal Fluid (CSF) | intraoperative
  BMS-986504 concentration will be quantified in CSF collected during Phase 0 surgery.
6-Month Progression Free Survival (PFS6) Rate | From date of Phase 0 surgery to date of disease recurrence or death, assessed over 27 months
  PFS6 rate of participants that had a positive PK response and enrolled into the Expansion Phase 1 component will be quantified.
Overall Survival (OS) | From date of surgery until death, due to any cause, assessed up to 27 months
  OS of participants that had a positive PK response and enrolled into the Expansion Phase 1 component will be summarized using Kaplan-Meier Curves and Estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Ivy Brain Tumor Center
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No